CLINICAL TRIAL: NCT01357746
Title: Detection, Estimation and Characterization of Pulmonary Blood Pressure by Transthoracic Parametric Doppler (TPD)
Brief Title: Measuring Blood Pressure in the Lung Circulation With Sonar Technology (Echo-Doppler)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Low recruitment
Sponsor: Echosense Ltd. (Industry)
Responsible Party: RACHEL SCHATZBERGER/CHIEF SCIENTIFIC OFFICER, Echosense Ltd.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: DOPO8
Record Dates: First submitted 2011-05-17; First posted 2011-05-23 (Estimated); Last update posted 2013-08-20 (Estimated); Status verified 2011-05

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: Pulmonary arterial blood pressure doppler
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Transthoracic pulmonary doppler recording — A 30 min recording of doppler signals from the right chest wall including measurements while the patient performs Valsalva maneuvers

SUMMARY:
This is a non-invasive study using a standard doppler echocardiographic transducer which records signals emanating from the lungs (TPD). These signals are caused by pulsation of blood vessels in the lung tissue.

The innovations in this study are:

1. The software processing of the reflected ultra-sound waves from the lung rendering a reproducible, clear and strong signal in sync with the cardiac cycle,
2. The observation based on pilot studies that blowing hard against resistance during recording (something called a Valsalva maneuver), affects the lung signal weakening it and even obliterating it as the pressure rises.

The investigators hypothesis is that since the signal comes from the blood vessels in the lung, the pressure at which the recorded signal disappears during the Valsalva maneuver represents the blood pressure in the lungs.

DETAILED DESCRIPTION:
Current methods for noninvasive measurement of pulmonary arterial blood pressure by standard echo-doppler equipment are fraught with uncertainty. So much so that patients being screened and followed for pulmonary arterial hypertension require right heart catheterization. An invasive and uncomfortable and potentially dangerous procedure.

This study is designed to confirm our preliminary observation that there is good correlation between Valsalva maneuver pressure and pulmonary arterial blood pressure.

Sixty patients undergoing right heart catheterization for clinical reasons will be studied.

The study itself is short, about 30 minutes, painless and done with the patient either sitting up in bed or semi-reclining. The probe is positioned over the right chest wall and the patient is requested to successively blow into a mouthpiece at rising pressures, to tolerance.

The results obtained using TPD to asses pulmonary arterial pressure will be compared to the results obtained at catheterization.

This is part of the development phase of the technology.

ELIGIBILITY:
Inclusion Criteria:

Eligibility

* Age 18 years or older
* Patients who are clinically suspected of having elevated pulmonary blood pressure , due to cardiac or cardio-pulmonary disease preferably any one or more of the conditions listed below, and due to have right heart catheterization as part of the diagnostic work-up:
* Patients with CHF
* Patients with primary pulmonary arterial hypertension
* Patients with COPD
* Patients with asthma
* Patients with interstitial lung disease
* Patients with sarcoidosis
* Signed informed consent.

Exclusion Criteria:

* Patients unable to cooperate.
* Inability to assume a sitting or supine position
* Patients with severe chest wall deformity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-07; Primary Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Reaching target enrollment number | 1-2 years
  Enrollment of 60 valid patients

SECONDARY OUTCOMES:
Lack of adverse effects | 1-2 years
  No adverse effects are expected but since this is a new application of old technolology safety is a possible issue.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Dragu, MD, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Department of Cardiology, Rambam Medical Center, Haifa, Israel